CLINICAL TRIAL: NCT02331966
Title: Molecular Pathways Involved in the Pathogenesis and Behavior of Mesenchymal Phosphaturic Tumors
Brief Title: Molecular Pathways Involved in the Pathogenesis and Behavior of Mesenchymal Phosphaturic Tumors Causing Oncogenic Osteomalacia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Maria Yavropoulou, Dr, AHEPA University Hospital
Other Study IDs: 51741
Record Dates: First submitted 2015-01-05; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Tumor Induced Oncogenic Osteomalacia
Keywords: FGF-23; GROWTH FACTORS RECEPTORS; RECURRENCES
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — RNA extraction from bone marrow and tissue samples from patients with tumor -induced osteomalacia
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The tumors that cause oncogenic osteomalacia (TIO) express and release in the circulation phosphaturic factors such as fibroblast growth factor-23 (FGF-23) that decrease renal phosphate absorption through acting in the proximal renal tubule and decreasing Type 2a and 2c sodium-phosphate co-transporter. They typically follow a benign clinical course and even in the rare malignant cases, local recurrence occurs in less than 5% and distant metastasis are very uncommon.

In this study we aim to investigate the role of other molecular pathways such as ERK1, ERK2, mTOR, EGFR, MEK1, MEK2, VEGFR3, AKT1, AKT2, IGFR-1, IGFR-2, PDGFRA, PDGFRB, cMET, FGFR2, apart from FGF23, KLOTHO and PHEX, in the behavior of histopathologically benign mesenchymal phosphaturic tumors.

DETAILED DESCRIPTION:
Study Protocol Cell Culture Bone marrow and tissue samples will be obtained from the patients after they will give their written informed consent. Material will be maintained in RPMI culture medium (Sigma, R0883, Germany). Peripheral blood mononuclear cells (PBMCs) from healthy donors will be used as control. For detection of cancer cells in our samples we perform flow cytometry using EpCAM magnetic beads (39-EPC-50; Gentaur), and the negative selection cells (non-cancerous) are isolated and then cultured in a 25-cm2 flask (5520100; Orange Scientific) with RPMI-1640 medium (R6504; Sigma).

Molecular analysis RNA is extracted from cell cultures using RNeasy Mini Kit (74105; Qiagen, Hilden; Germany). iScript cDNA synthesis kit (1708891; Bio-Rad, CA; USA), is used for cDNA synthesis and Real-time polymerase chain reaction (PCR), is performed using the iTaq Universal SYBR Green Supermix (1725124; Bio-Rad). Specific primers for each marker and for an endogenous control gene (18S rRNA) is designed using Genamic Expression 1.1 software. A universal Reference RNA consisting of 10 human cancer cell lines (740000-41; Agilent) as well as human genomic DNA (G304A; Promega) will be used in quantitative PCR (qPCR) reactions Statistical analysis The qPCR results will be tested according to the Kolmogorov-Smirnov test; All the reactions (molecular assays, flow cytometry) are performed in triplicates. A p value <0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

Patients with tumor induced osteomalacia

Exclusion Criteria:

None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with tumor induced osteomalacia
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Differential expression of Molecular pathways in tumors inducing oncogenic osteomalacia | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Maria P. Yavropoulou, M.D, Principal Investigator — AHEPA University Hospital
Locations (1):
- 1st Department of Internal Medicine AHEPA University Hospital, Thessaloniki, Greece